CLINICAL TRIAL: NCT03532542
Title: Long-term, Open-label Extension Study for Patients With Duchenne Muscular Dystrophy Enrolled in Clinical Trials Evaluating Casimersen or Golodirsen
Brief Title: An Extension Study to Evaluate Casimersen or Golodirsen in Patients With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was stopped to reduce the clinical trial burden on participants while ensuring continued treatment via a post-trial access program with commercially available casimersen and golodirsen. Study was not terminated due to safety concerns.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4045-302; 2017-004625-32 (EudraCT Number)
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Exon Skipping; DMD; Exon 53; Exon 45; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — casimersen; golodirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Casimersen (Experimental): Patients amenable to exon 45 skipping who have completed a clinical trial evaluating casimersen will receive open-label casimersen intravenous (IV) infusions, weekly, at 30 mg/kg for up to 144 Weeks.
  Interventions: Drug: Casimersen
- Golodirsen (Experimental): Patients amenable to exon 53 skipping who have completed a clinical trial evaluating golodirsen will receive open-label golodirsen intravenous (IV) infusions, weekly, at 30 mg/kg for up to 144 Weeks.
  Interventions: Drug: Golodirsen

INTERVENTIONS:
Drug: Casimersen — Casimersen solution for IV infusion
  Other Names: SRP-4045; AMONDYS 45
  Arms: Casimersen
Drug: Golodirsen — Golodirsen solution for IV infusion
  Other Names: SRP-4053; VYONDYS 53
  Arms: Golodirsen

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of long-term treatment with casimersen or golodirsen in patients with Duchenne muscular dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

* Completed a clinical trial evaluating casimersen or golodirsen, per protocol.
* Is between 7 and 23 years of age, inclusive, at enrollment.

Other inclusion/exclusion criteria apply.

Ages: 7 Years to 23 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 171 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (50):
- United States (25):
  - Neuromuscular Research Center, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Rady Children's Hospital- San Diego, San Diego, California
  - UF Health: University of Florida Clinical Research Center, Gainesville, Florida
  - NW Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - University of Iowa Childrens Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Las Vegas Clinic, Las Vegas, Nevada
  - University of Rochester Medical Center - Department of Neurology, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Abigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospital for Children, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah - PPDS, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital of Wisconsin, Corporate Center Suite 540, Milwaukee, Wisconsin
- Belgium (2):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven
- University Multiprofile Hospital for active treatment Aleksandrovska EAD Clinic of Neurological Diseases, Sofia, Bulgaria
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- Czechia (2):
  - Fakultni nemocnice Brno, Klinika detske neurologie LF MU a FN Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- France (2):
  - Hotel Dieu- CHU Nantes, Nantes
  - Hôpital Armand Trousseau, Paris
- Germany (2):
  - Universitatsklinikum Freiberg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Italy (3):
  - UOSD Centro Traslazionale di Miologia e Patologie Neurogenerative, Genoa, Liguria
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant' Anna, Cona
  - Fondazione Policlinico Universitario A Gemelli, Milan
- Poland (2):
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Klinica Neurologii Rozwojowej, Gdansk
- Spain (3):
  - Hospital de La Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Provningsenhet Barn, Drottning Silvias Och Ungdomssjukhus, Gothenburg, Sweden
- United Kingdom (4):
  - Leeds General Infirmary, Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital (GOSH), London
  - Royal Victoria Infirmary, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants amenable to exon 53 or exon 45 skipping were enrolled into this study from Study 4045-101 (NCT02530905), Study 4053-101 (NCT02310906), and Study 4045-301 (NCT02500381).
Groups:
- Golodirsen: Participants amenable to exon 53 skipping who have completed a clinical trial evaluating golodirsen received open-label golodirsen intravenous (IV) infusions, weekly, at 30 milligrams/kilogram (mg/kg) for up to 144 weeks.
- Casimersen: Participants amenable to exon 45 skipping who have completed a clinical trial evaluating casimersen received open-label casimersen IV infusions, weekly, at 30 mg/kg for up to 144 weeks.
Period: Overall Study
Arm/Group | Golodirsen | Casimersen
Started | 74 | 97
Received at Least 1 Dose of Study Drug (Safety Analysis Set) | 74 | 97
Completed | 26 | 27
Not Completed | 48 | 70
Not completed — Death | 1 | 0
Not completed — Study Terminated by Sponsor | 41 | 65
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study drug (golodirsen or casimersen).
Groups:
- Golodirsen: Participants amenable to exon 53 skipping who have completed a clinical trial evaluating golodirsen received open-label golodirsen IV infusions, weekly, at 30 mg/kg for up to 144 weeks.
- Total: Total of all reporting groups
Arm/Group | Golodirsen | Casimersen | Total
Number analyzed (Participants) | 74 | 97 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (2.14) | 12.2 (2.57) | 12.0 (2.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 74 | 97 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 54 | 89 | 143
  Unknown or Not Reported | 10 | 2 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 65 | 86 | 151
  Black | 1 | 0 | 1
  Asian | 4 | 7 | 11
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: A treatment-emergent adverse event (TEAE) was any untoward medical occurrence in a clinical study participant that did not necessarily have a causal relationship with the study drug. A TEAE could, therefore, be any unfavorable and unintended symptom, sign, disease, condition, or test abnormality that occurred during or after administration of the study drug, whether or not considered related to the study drug. A TESAE was any TEAE that resulted in any of the following outcomes: death, a life-threatening event, required or prolonged inpatient hospitalization, persistent or significant disability/incapacity, or an important medical event (that is, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the previously mentioned outcomes). A summary of serious and all other non-serious TEAEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 33 days after the last infusion of study drug (up to approximately 149 weeks)
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of study drug (golodirsen or casimersen).
Measure: Count of Participants; unit: Participants
Arm/Group | Golodirsen | Casimersen
Number analyzed (Participants) | 74 | 97
Participants | 12 | 22

ADVERSE EVENTS:
Time Frame: Up to 33 days after the last infusion of study drug (up to approximately 149 weeks)
Description: All reported adverse event data based upon Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug (golodirsen or casimersen).
Arm/Group | Golodirsen | Casimersen
All-Cause Mortality (participants affected / at risk) | 1/74 | 0/97
Serious Adverse Events (participants affected / at risk) | 12/74 | 22/97
Other Adverse Events (participants affected / at risk) | 63/74 | 93/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golodirsen (N=74) | Casimersen (N=97)
Femur fracture (Injury, poisoning and procedural complications) | 3 | 8
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal embolism (Renal and urinary disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuromuscular scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Distributive shock (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Golodirsen (N=74) | Casimersen (N=97)
COVID-19 (Infections and infestations) | 10 | 27
Nasopharyngitis (Infections and infestations) | 26 | 21
Upper respiratory tract infection (Infections and infestations) | 7 | 15
Influenza (Infections and infestations) | 6 | 7
Gastroenteritis (Infections and infestations) | 5 | 6
Rhinitis (Infections and infestations) | 8 | 6
Fall (Injury, poisoning and procedural complications) | 19 | 17
Contusion (Injury, poisoning and procedural complications) | 8 | 13
Back injury (Injury, poisoning and procedural complications) | 3 | 9
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 7
Femur fracture (Injury, poisoning and procedural complications) | 5 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 9 | 5
Limb injury (Injury, poisoning and procedural complications) | 6 | 4
Joint injury (Injury, poisoning and procedural complications) | 5 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 13
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 22 | 15
Diarrhoea (Gastrointestinal disorders) | 13 | 11
Constipation (Gastrointestinal disorders) | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 7 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Pyrexia (General disorders) | 13 | 22
Pain (General disorders) | 2 | 6
Adverse drug reaction (General disorders) | 3 | 5
Gait inability (General disorders) | 5 | 1
Headache (Nervous system disorders) | 22 | 25
Dizziness (Nervous system disorders) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 8
Ingrowing nail (Skin and subcutaneous tissue disorders) | 4 | 3
Urine protein/creatinine ratio increased (Investigations) | 7 | 8
Haematuria (Renal and urinary disorders) | 6 | 5
Proteinuria (Renal and urinary disorders) | 4 | 2
Cataract (Eye disorders) | 6 | 5
Haematoma (Vascular disorders) | 4 | 4

LIMITATIONS AND CAVEATS:
This study was terminated before all participants had reached the last protocol-defined end-of-study visit. Study termination resulted in participants either being transitioned to a post-trial access program, to another study, or they declined further treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03532542/Prot_000.pdf